CLINICAL TRIAL: NCT07043322
Title: Clinical Study to Evaluate Efficacy of Cabergoline to Coasting in Reducing the Incidence of Ovarian Hyperstimulation Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 874
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Group 1 (coasting only): In their ICSI cycle patients will take 0.25 mg of cabergoline daily for 8 days from HCG triggering day to prevent OHSS. Early OHSS is assessed at day of embryo transfer and 7 days after this date. Late OHSS is assessed 14 days after embryo transfer.
  Interventions: Procedure: Coasting
- Cabergoline group (Active Comparator): Coasting plus cabergoline: In their ICSI cycle patients will continue their agonist treatment while stopping the human menopausal gonadotropin (hMG) injections for 1 day plus receiving 0.25 mg of cabergoline daily for 8 days from HCG triggering day to prevent OHSS. Early OHSS is assessed at day of embryo transfer and 7 days after this date. Late OHSS is assessed 14 days after embryo transfer.
  Interventions: Procedure: Coasting; Drug: Cabergoline

INTERVENTIONS:
Procedure: Coasting — In their ICSI cycle patients will continue their agonist treatment while stopping the human menopausal gonadotropin (hMG) injections for 1 to 3 days until drop of estradiol to a safe level to prevent OHSS. Early OHSS is assessed at day of embryo transfer and 7 days after this date. Late OHSS is assessed 14 days after embryo transfer.
Drug: Cabergoline — Cabergoline is used to treat different types of medical problems that occur when too much of the hormone prolactin is produced. It can be used to treat certain menstrual problems, fertility problems in men and women, and pituitary prolactinomas
  Arms: Cabergoline group

SUMMARY:
Ovarian hyperstimulation syndrome (OHSS) is a serious iatrogenic complication of controlled ovarian stimulation of gonadotrophin-Stimulated ovarian cycles. It is theorized to manifest systemically as a result of vasoactive mediators like vascular endothelium growth factor (VEGF) being released from hyperstimulated ovaries. As a result, capillary permeability is increased which causes the extravasation of fluid from the intravascular compartment into the third space. The haemoconcentration which ensues results in complications such as hypercoagulability and reduced end organ perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-38 years
* Body mass index (calculated as weight in kilograms divided by the square of height in meters) < 30 kg/m2.
* A long luteal protocol is used for ovarian stimulation.
* Day 2 FSH <10 mIU/L and E2< 50 pg/ml
* High risk of OHSS, defined as having more than 20 follicles >12 mm in diameter and/or E2 levels > 3000 pg/ml when the size of the leading follicle is > 15 mm

Exclusion Criteria:

The presence of chronic medical diseases, including liver cell failure, renal failure, uncontrolled hypertension, uncontrolled diabetes mellitus, or class 3 or 4 function heart disease in the New York heart association classification.

Allergy to Cabergoline.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Occurrence and severity of OHSS | 1 month
  The primary outcome of this study is the occurrence and severity of OHSS. OHSS was defined as abdominal pain and distention associated with nausea and vomiting and ovarian enlargement > 8 cm. The severity of OHSS will be assessed (mild, moderate, severe, and clinical) according to the American Society for Reproductive Medicine guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa Bahaa, Damietta, New Damietta, Egypt